CLINICAL TRIAL: NCT04536337
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, First-in-Human Study of Orally Administered ALG-000184 to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single-Ascending Doses (Part 1) and Multiple-Ascending Doses in Healthy Volunteers (Part 2), and Multiple Doses in Subjects With Chronic Hepatitis B (Part 3)
Brief Title: A Study of ALG-000184 Drug to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Single and Multiple Doses in Healthy Volunteers and CHB Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALG-000184-201
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Intervention Model Description: This is a parallel-group study with several parts. In Parts 1-3, participants are randomized in a 4:1 ratio to receive either ALG-000184 or matching placebo. In Part 4, participants are randomized in a 4:1 ratio to receive either ALG-000184 plus entecavir or placebo plus entecavir. In Part 5, all participants receive open-label ALG-000184 plus entecavir.
  The study follows a dose-escalation design where doses are increased across cohorts based on safety and pharmacokinetic data from previous cohorts. Each participant remains in their assigned treatment group throughout their participation in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ALG-000184 (Experimental): Oral tablet(s) of ALG-000184 in HV or CHB subjects once daily for up to 96 weeks
  Interventions: Drug: ALG-000184
- Placebo (Placebo Comparator): Oral tablet(s) of placebo in HV or CHB subjects once daily for up to 12 weeks
  Interventions: Drug: Placebo
- Entecavir in combination with ALG-000184 (Active Comparator): Oral tablet(s) of ALG-000184 in combination with Entecavir in CHB subjects once or twice daily for up to 96 weeks
  Interventions: Drug: ALG-000184; Drug: Entecavir
- Placebo plus Entecavir (Active Comparator): Oral tablet(s) of matching placebo in combination with Entecavir in CHB subjects once daily for 12 weeks, with option to switch to open-label ALG-000184 plus Entecavir for up to 96 weeks (Part 4).
  Interventions: Drug: ALG-000184; Drug: Entecavir
- Open-label ALG-000184 plus Entecavir (Experimental): Open-label oral tablet(s) of ALG-000184 in combination with Entecavir in CHB subjects once daily for up to 96 weeks (Part 5)
  Interventions: Drug: Placebo; Drug: Entecavir

INTERVENTIONS:
Drug: ALG-000184 — Single or multiple doses of ALG-000184
  Arms: ALG-000184; Entecavir in combination with ALG-000184; Placebo plus Entecavir
Drug: Placebo — Single or multiple doses of Placebo
  Arms: Open-label ALG-000184 plus Entecavir; Placebo
Drug: Entecavir — multiple doses of Entecavir
  Arms: Entecavir in combination with ALG-000184; Open-label ALG-000184 plus Entecavir; Placebo plus Entecavir

SUMMARY:
The goal of this clinical trial is to learn if ALG-000184 is safe, well-tolerated, and works to treat chronic hepatitis B virus (HBV) infection. The main questions it aims to answer are:

Is ALG-000184 safe and well-tolerated when given alone or with entecavir (a standard HBV treatment)? Does ALG-000184 reduce HBV viral levels in the blood of patients with chronic hepatitis B? How does the body process ALG-000184 (pharmacokinetics)?

Researchers will compare ALG-000184 to placebo (a look-alike substance that contains no drug) to see if ALG-000184 works better at reducing hepatitis B viral markers.

The study has five parts:

Parts 1 and 2: Healthy volunteers will receive single or multiple doses of ALG-000184 or placebo Part 3: Patients with chronic hepatitis B will receive ALG-000184 or placebo daily for 28 days Part 4: Patients with chronic hepatitis B will receive ALG-000184 or placebo combined with entecavir for 12 weeks (may be extended up to 96 weeks) Part 5: Additional groups of patients with chronic hepatitis B will receive ALG-000184 with entecavir for 12 weeks (may be extended up to 96 weeks)

Participants will:

Take study medication orally as directed Visit the clinic regularly for blood tests, physical examinations, and other safety assessments Have their HBV viral markers measured to determine if the treatment is working

DETAILED DESCRIPTION:
ALG-000184-201 is a Phase 1, double-blind, randomized, placebo-controlled study evaluating ALG-000184, a novel capsid assembly modulator (CAM) targeting hepatitis B virus (HBV).

ALG-000184 is a prodrug that is converted to ALG-001075, a Class E CAM that inhibits HBV replication through two mechanisms: (1) blocking pregenomic RNA encapsidation, and (2) preventing the formation and transcription of covalently closed circular DNA (cccDNA).

The study employs a sequential approach, beginning with single-ascending dose (SAD) and multiple-ascending dose (MAD) evaluations in healthy volunteers, then progressing to monotherapy assessments in chronic hepatitis B (CHB) subjects, and finally testing combination therapy with entecavir.

A Study Review Committee (SRC) oversees safety throughout the trial and determines dose escalation based on predefined criteria. Each cohort in Parts 1-3 includes a 4:1 (ALG-000184:placebo) randomization ratio, while Parts 4-5 include extended treatment durations to evaluate longer-term efficacy and safety.

The study includes comprehensive pharmacokinetic assessments and extensive virologic evaluations (HBV DNA, HBV RNA, HBsAg, HBeAg, HBcrAg, and resistance monitoring). An ALT Flare Committee specifically reviews and manages liver-related safety events.

Part 4 focuses on HBeAg-positive subjects to explore potential HBsAg declines, as the secondary mechanism of action of ALG-000184 may be more pronounced in subjects with higher cccDNA levels. The trial includes provisions for extending treatment duration up to 96 weeks based on emerging safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria for All Subjects:

1. Female subjects must have a negative serum pregnancy test at screening
2. Subjects must have a 12-lead electrocardiogram (ECG) that meets the protocol criteria

   Inclusion Criteria for Healthy Volunteers:

   In addition to inclusion criteria 1-2, the following inclusion criteria also apply to HV's (Parts 1 and 2)
3. Male or female between 18 and 55 years of age, extremes included.
4. Subjects must have a body mass index (BMI; weight in kg divided by the square of height in meters) of 18.0 to 32.0 kg/m2, extremes included.

CHB Subjects:

In addition to inclusion criteria 1-4, the following inclusion criteria also apply to CHB subjects:

All of the Following criteria apply to Part 3 at screening:

5 .Subjects must be 18 to 65 years of age, extremes included.

6.CHB subjects must have a BMI of 18.0 to 35.0 kg/m2, extremes included.

7.CHB subjects who at screening, have not received treatment with an approved or investigational medicine, or have never received treatment with HBV antiviral medicines

All of the following criteria apply to Part 4 Cohorts A & B, unless otherwise specified, at Screening:

8.Subjects must be 18 to 65 years of age, extremes included.

9.Subjects must have a BMI of 18.0 to 35.0 kg/m2, extremes included

10.Subjects must be HBeAg positive (HBeAg ≥LLOQ and HBeAb negative)

11.Subjects enrolled in Part 4 Cohort A and B must have a history of Chronic Hepatitis B

12. Subjects must have ALT and AST must have ≤1.2×ULN or ≤5×ULN

All of the following criteria apply to Part 5 at Screening

13.Subjects must be 18 to 65 years of age, extremes included.

14. Subjects have a BMI of 17.0 to 35.0 kg/m2, extremes included

15.Subjects could belong to any of the following treatment categories: treatment naïve (TN), currently not treated (CNT) , virologically suppressed.

Exclusion Criteria

Exclusion Criteria for All Subjects:

1. Subjects with any previous or current illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject, or pose an additional risk in administering study drug to the subject, or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT syndrome, or history of clinical evidence at screening of significant or unstable cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Subject with a current history of clinically significant (as determined by investigator) skin disease requiring intermittent or chronic treatment
5. Excessive use of alcohol, defined as regular consumption of ≥14 standard drinks/week for women and ≥21 standard drinks/week for men
6. Subjects with Hepatitis A, B, C, D, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection

   Exclusion Criteria for Healthy Volunteers (Parts 1 and 2):

   In addition to exclusion criteria 1-6, the following exclusion criteria also apply to HV's (Parts 1 and 2)
7. Unwilling to abstain from alcohol use for 48 hours prior to start of dosing through end of study follow up.
8. Positive alcohol or cotinine test at screening and Day -1.
9. Subjects with renal dysfunction (e.g., estimated creatinine clearance <90 mL/min/1.73 m2at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula).

   Exclusion Criteria for CHB Subjects (Parts 3, 4, and 5):

   All exclusion criteria listed above for healthy volunteers apply also to CHB subjects, except for exclusion Criteria 9 (requirement relative to cotinine).All the following exclusion criteria apply to Parts 3, 4, and 5, unless otherwise specified.
10. Subjects who are positive for anti-HBs antibodies.
11. For HBeAg-positive subjects, they should be negative for anti-HBe antibodies (Parts 4 and 5)
12. Subject with any history or current evidence of hepatic decompensation such as: variceal bleeding, spontaneous bacterial peritonitis, ascites, hepatic encephalopathy, or active jaundice (within the last year).
13. History or current evidence of cirrhosis.
14. Subjects with liver fibrosis that is classified as Metavir Score ≥F3 liver disease
15. Subjects with signs of hepatocellular carcinoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 8 days for Part 1
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 21 days for Part 2
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | up to 112 days for Part 3
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 756 days for parts 4 & 5
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1 of ALG-184 in combination with Entecavir (Parts 4 and 5)

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | Predose up to763 Days
  Pharmacokinetic parameters of ALG-000184 in plasma
Area under the concentration time curve [AUC] | Predose up to 763 Days
  Pharmacokinetic parameters of ALG-000184 in plasma
Time to maximum plasma concentration [Tmax] | Predose up to 763 Days
  pharmacokinetic parameters of ALG-000184 in plasma
Half-time [t1/2] | Predose up to 763 Days
  Pharmacokinetic parameters of ALG-000184 in plasma
Minimum Plasma Concentration [Cmin] | Predose up to 763 Days
  Pharmacokinetic parameters of ALG-000184 in plasma
Change in HBV DNA from baseline through Day 812 in Multiple Dose HBV Infected Patients | Screening up to Day 812

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (2):
  - Saint Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Western Health, Footscray, Victoria
- China (3):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Hospital of Jilin University, Changchun, Jilin
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales, Shatin
- CAP Research, Quatre Bornes, Mauritius, Mauritius
- PMSI Republican Clinical Hospital "T. Mosneaga", ARENSIA Exploratory Medicine Phase I Unit, Chisinau, Moldova
- ACS, Auckland, New Zealand

REFERENCES:
- [Derived] Yuen MF, Agarwal K, Jucov A, Hou J, Niu J, Ding Y, Haceatrean A, Liang X, Xu J, Wu M, Le K, Lin TI, Blatt L, Chanda S, Fry J, Gane E. ALG-000184 (pevifoscorvir sodium) monotherapy in participants with chronic HBV infection: a phase 1, multicentre, randomised, dose escalation trial. Lancet Gastroenterol Hepatol. 2026 Jan 16:S2468-1253(25)00293-6. doi: 10.1016/S2468-1253(25)00293-6. Online ahead of print. PMID 41554267
- [Derived] Gane E, Schwabe C, Wu M, Lin TI, Blatt L, Fry J, Chanda S, Le K. A Phase 1 study of the safety, tolerability, and pharmacokinetics of ALG-000184 (pevifoscorvir sodium), a novel Class E capsid assembly modulator, in healthy participants. Antivir Ther. 2025 Dec;30(6):13596535251392955. doi: 10.1177/13596535251392955. Epub 2025 Nov 21. PMID 41268712
- [Derived] Li C, Wu M, Zhang H, Mai J, Yang L, Ding Y, Niu J, Mao J, Wu W, Zhang D, Tang Y, Yan W. Safety, Tolerability, and Pharmacokinetics of the Novel Hepatitis B Virus Capsid Assembly Modulator GST-HG141 in Healthy Chinese Subjects: a First-in-Human Single- and Multiple-Dose Escalation Trial. Antimicrob Agents Chemother. 2021 Sep 17;65(10):e0122021. doi: 10.1128/AAC.01220-21. Epub 2021 Jul 19. PMID 34280012